CLINICAL TRIAL: NCT05483634
Title: Compare the Effectiveness and Side Effects of Vaginal Estrogen and Platelet-rich Plasma Over Women With Genitourinary Syndrome of Menopause
Brief Title: Compare Vaginal Estrogen and Platelet-rich Plasma Over Women With Genitourinary Syndrome of Menopause
Status: Not yet recruiting | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hui-Hsuan Lau, MD, Doctor, Mackay Memorial Hospital
Other Study IDs: 19MMHIS340e
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Menopause; Platelet-rich Plasma; Estrogen Replacement Therapy; Vaginal Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Genital urinary symptoms of menopause: Menopause for one year, or age above 45 with symptoms of GSM
  Interventions: Drug: Vaginal estrogen supplement; Procedure: Platelet-rich plasma injection

INTERVENTIONS:
Drug: Vaginal estrogen supplement — Daily vaginal estrogen supplement, then twice per week. Continue for three months.
Procedure: Platelet-rich plasma injection — Monthly platelet-rich plasma injection for three months

SUMMARY:
The definition of Genitourinary Syndrome of Menopause (GSM) is the decline of estrogens during menopause results in symptoms and clinical signs from both systems. Estrogen and other hormones production decrease after menopause because the ovaries lose their effectiveness, leading to mucosal atrophy, reduced vaginal moisture, dysuria, urgency, recurrent infection, burning, pruritus and dyspareunia.

The treatment included vaginal estrogen supplement, vaginal hyaluronic acid supplement, vaginal laser, platelet rich plasma, etc. Observational cohort study will be used for study design, and questionnaire, pelvic examination, vaginal pap smear with maturation index (MI), vaginal pH, and other methods will be used for evaluation of the effectiveness and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Women with menopause
* Patients with symptoms of genitourinary syndrome of menopause

Exclusion Criteria:

* Genitourinary bleeding or infection without definitive diagnosis
* Coagulopathy
* Allergy to medication or therapy related with the treatment
* Chronic disease that might influence outcome
* Using medication that might influence outcome in 30 days
* Using hormone or steroid within 8 weeks

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Menopause for one year Age above 45 with symptoms of GSM
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 2022/8/10-2024/2/28
  Changes in GSM symptoms include vaginal dryness, dyspareunia, itching, burning, dysuria
Vaginal health index score (VHIS) | 2022/8/10-2024/2/28
  One of the most commonly used scores for the evaluation of vaginal elasticity, secretions, pH, the presence of petechiae on the epithelial mucosa, and hydration
Female Sexual Function Index (FSFI) | 2022/8/10-2024/2/28
  A brief multidimensional scale for assessing sexual function in women.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsuan Lau, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gandhi J, Chen A, Dagur G, Suh Y, Smith N, Cali B, Khan SA. Genitourinary syndrome of menopause: an overview of clinical manifestations, pathophysiology, etiology, evaluation, and management. Am J Obstet Gynecol. 2016 Dec;215(6):704-711. doi: 10.1016/j.ajog.2016.07.045. Epub 2016 Jul 26. PMID 27472999
- [Background] Pitsouni E, Grigoriadis T, Falagas ME, Salvatore S, Athanasiou S. Laser therapy for the genitourinary syndrome of menopause. A systematic review and meta-analysis. Maturitas. 2017 Sep;103:78-88. doi: 10.1016/j.maturitas.2017.06.029. Epub 2017 Jun 27. PMID 28778337
- [Background] Pitsouni E, Grigoriadis T, Douskos A, Kyriakidou M, Falagas ME, Athanasiou S. Efficacy of vaginal therapies alternative to vaginal estrogens on sexual function and orgasm of menopausal women: A systematic review and meta-analysis of randomized controlled trials. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:45-56. doi: 10.1016/j.ejogrb.2018.08.008. Epub 2018 Aug 6. PMID 30103082
- [Background] Najjarzadeh M, Mohammad Alizadeh Charandabi S, Mohammadi M, Mirghafourvand M. Comparison of the effect of hyaluronic acid and estrogen on atrophic vaginitis in menopausal women: A systematic review. Post Reprod Health. 2019 Jun;25(2):100-108. doi: 10.1177/2053369119830818. Epub 2019 Feb 24. No abstract available. PMID 30798700
- [Background] Saleh DM, Abdelghani R. Clinical evaluation of autologous platelet rich plasma injection in postmenopausal vulvovaginal atrophy: A pilot study. J Cosmet Dermatol. 2022 Oct;21(10):4269-4275. doi: 10.1111/jocd.14873. Epub 2022 Mar 7. PMID 35194935